CLINICAL TRIAL: NCT04476225
Title: Induced Pluripotent Stem Cells for Disease Research
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 19-27665
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Hirschsprung Disease
Keywords: Hirschsprung Disease
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with Hirschsprung Disease: Individuals with Hirschsprung disease
- Unaffected Relatives: Unaffected relatives of individuals with Hirschsprung disease

SUMMARY:
The aim of this study is to determine the contribution of genetic factors to the pathogenesis of diseases, including diseases such as Parkinson's disease, Hirschsprung's disease, and autism. Patient-derived cellular models of diseases will be developed, which will require the collection of blood samples from patients and healthy individuals in order to generate induced pluripotent stem cells (iPSCs) for the development of iPSC-derived human cell cultures. These human cellular models will be phenotyped using a variety of methods, including cellular, molecular, and biochemical assays. Because these human cellular models will retain the genetic background from the patients and control subjects, this will allow us to determine the contribution of genetics to disease phenotypes. Such disease-specific pluripotent stem cell lines will be invaluable tools for many basic and translational research applications, including pathophysiological studies in a developmental context, and innovation and screening of small molecule drugs capable of reversing the disease phenotype and potentially leading to a cure for a broad range of diseases, where appropriate in vitro or in vivo disease models do not exist.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with Hirschsprung disease
* Any disease severity accepted
* Individuals with or without other health issues accepted
* Unaffected / healthy relatives of individuals with Hirschsprung disease

Exclusion Criteria:

* Individuals who are unwilling or unable to provide blood sample
* Individuals who are unwilling or unable to provide informed consent
* Individuals who are outside the age range permitted for our study will be excluded. Our study will only perform blood draws from individuals ages 13 and above.

Ages: 13 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with Hirschsprung disease and their unaffacted family members
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
Whole blood sample collection | 52 weeks after sample collection
  Collect human peripheral blood mononuclear cells (PBMCs) and reprogram into iPSCs.
iPSC disease modeling | 200 weeks after sample collection
  Use patient-derived iPSCs to develop models of human diseases and to determine the contribution of patient genetic factors to disease pathogenesis

CONTACTS AND LOCATIONS:
Overall Officials: Steve Finkbeiner, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No